CLINICAL TRIAL: NCT00381277
Title: The Effects of Sports Drinks on Urinary Lithogenicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: David S Goldfarb MD, New York Harbor VA Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DG-1
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Urolithiasis
Keywords: nephrolithiasis; citrate; oxalate
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis | interventions — gatorade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gatorade
Drug: Performance

SUMMARY:
The effect of sports drinks on the tendency to form kidney stones has not been assessed. Patients will drink 1 liter a day of 2 sports drinks and collect urine to determine changes in urine chemistry that may decrease the risk of forming stones.

DETAILED DESCRIPTION:
Participants will drink 1 liter of water each day for one week in the control period, then 1 liter of sports drink each day for one week during the experimental period. Urine collections will be performed during both periods. Diet will be chosen by participants and a food diary will be kept so that participants can replicate diet during the urine collections.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old
* men and women
* able to sign informed consent

Exclusion Criteria:

* history of kidney stones
* bone disease
* parathyroid disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-03; Primary Completion 2006-03 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Urinary supersaturation of calcium oxalate
Urinary citrate excretion
Urinary calcium excretion
Urinary sodium excretion

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldfarb, MD, Study Director — New York Harbor VAMC
Locations (1):
- New York Harbor VAMC, New York, New York, United States